CLINICAL TRIAL: NCT00267293
Title: Ibuprofen Alone and in Combination With Acetaminophen for Treatment of Fever
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Children Youth and Family Consortium (Other)
Responsible Party: Principal Investigator, Ian M. Paul, M.D., M.Sc., Professor of Pediatrics and Public Health Sciences, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HY03-127
Record Dates: First submitted 2005-12-16; First posted 2005-12-20 (Estimated); Results first posted 2012-05-09 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Fever
Keywords: fever treatment; children
MeSH Terms: conditions — Fever | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): At time 0 child is given an appropriate dose of Ibuprofen (10mg/kg)
  Interventions: Drug: Ibuprofen
- B (Experimental): At time 0 child is given an appropriate dose of Ibuprofen (10mg/kg) and an appropriate dose of Acetaminophen (15 mg/kg)
  Interventions: Drug: Acetaminophen; Drug: Ibuprofen
- C (Experimental): At time 0 child is given an appropriate dose of Ibuprofen (10mg/kg) and at time 3 hours is given an appropriate dose of Acetaminophen (15 mg/kg)
  Interventions: Drug: Acetaminophen; Drug: Ibuprofen

INTERVENTIONS:
Drug: Acetaminophen — Given for fever control 15mg/kg
  Arms: B; C
Drug: Ibuprofen — Given for fever control 10 mg/kg

SUMMARY:
Currently, when a child has fever either ibuprofen (e.g. Motrin, Advil) or acetaminophen (e.g. Tylenol) is given. Both Ibuprofen and Acetaminophen are approved for over the counter use for treatment of fever by the Food and Drug Administration (FDA). This study hopes to determine whether giving both medications together is better than giving one medication alone for the treatment of fever.

DETAILED DESCRIPTION:
Despite a lack of evidence to support their fears, a majority of parents, pediatricians, and pediatric nurses believe that fever can be dangerous to a child. This "fever phobia" has caused a majority of caregivers to aggressively treat fever with antipyretics such as ibuprofen and acetaminophen, often in combination. Although there is scant data to support the use of these medications together for fever control and none using alternating regimens, it was recently reported that 50% of pediatricians and 70% of pediatricians with less than 5 years of experience advise parents to alternate acetaminophen and ibuprofen as an attempt to achieve maximal antipyresis. While a combination of aspirin (no longer used for antipyresis in children) and acetaminophen has been shown to be superior to either agent alone for fever reduction, these data cannot be extrapolated to the pairing of ibuprofen and acetaminophen.

There is evidence that combinations of acetaminophen and non-steroidal anti-inflammatory drugs (NSAIDs) are more effective for the treatment of pain and can reduce opioid use when compared with a single agent. Improved activity and alertness in children have been reported after antipyretic administration.

It is believed that acetaminophen and ibuprofen may be safely used together because the two medications have significantly different pathways of metabolism that are not affected by each other, and have been used abroad in combination form for over a decade. Both acetaminophen and ibuprofen have been shown to be safe when given individually or together in recommended doses for short term use. There are no reports of adverse effects from combination therapy with standard doses.

In addition, while it now appears that fever itself is probably a protective physiologic response, under different circumstances it has the potential to be harmful. Fever increases the metabolic rate approximately 10% for every 1 degree C rise in body temperature. The myocardial depression,orthostatic dysfunction, and increases in oxygen consumption, respiratory minute volume, and respiratory quotient that occur may not be tolerated by all patients including some children.

Because of the ubiquitous nature of the problem, childhood fever, this study has the potential to immediately impact the way clinicians and parents treat children with fever. If the combination regimens are not shown to be superior, it could limit improper medication administration and overdose. If it is superior, the combination of medications may improve other symptoms associated with fever such as discomfort. Either way, it will fill the gap that exists in the evidence-based approach to the management of childhood fever and immediately impact current practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months - 7 years of age at time of the fever.
* Initial temperature of 38.0C (100.4F) or more.
* Ability to cooperate with serial temporal artery temperature measurements.
* Ability to take medications by mouth.
* Willingness of the child's guardian/sponsor to give informed consent

Exclusion Criteria:

* Patients who have received acetaminophen within 6 hours of presentation, or ibuprofen, aspirin, or other non-steroidal anti-inflammatory medications within 8 hours of presentation.
* Patients >=3 years of age that have received narcotics in the previous 24 hours.
* Children with weight >60 kg. Treatment of children with weights >60 kg will result in greater than recommended adult doses of the medications.
* History of adverse reaction to any study medication ingredient.
* History of diabetes mellitis, renal dysfunction, hepatic dysfunction, or thrombocytopenia.
* Presence of moderate or severe dehydration.
* Inclusion in the trial on 3 previous occasions
* Medical judgment that the severity of the underlying illness prohibits inclusion.

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2006-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian M Paul, MD, Principal Investigator — Penn State Milton S. Hershey Children's Hospital
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Paul IM, Sturgis SA, Yang C, Engle L, Watts H, Berlin CM Jr. Efficacy of standard doses of Ibuprofen alone, alternating, and combined with acetaminophen for the treatment of febrile children. Clin Ther. 2010 Dec;32(14):2433-40. doi: 10.1016/j.clinthera.2011.01.006. PMID 21353111
- See also: Penn State Milton S. Hershey Children's Hospital Pediatric Clinical Research Office — http://www.hmc.psu.edu/pedsclinicalresearch/index.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Ibuprofen Alone: Time 0 Ibuprofen (10mg/kg)given. Temperature in °C measured hourly for 6 hours.
- Group B: Ibuprofen and Acetaminophen: time 0 child Ibuprofen (10mg/kg) and Acetaminophen (15 mg/kg)given. Temperature in °C measured hourly for 6 hours.
- Group C: Ibuprofen Then Acetaminophen: Time 0 child is given Ibuprofen (10mg/kg) and at time 3 hours is given (15 mg/kg. Temperature in °C measured hourly for 6 hours.
Period: Overall Study
Arm/Group | Group A: Ibuprofen Alone | Group B: Ibuprofen and Acetaminophen | Group C: Ibuprofen Then Acetaminophen
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Ibuprofen Alone | Group B: Ibuprofen and Acetaminophen | Group C: Ibuprofen Then Acetaminophen | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 20 | 20 | 60
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 3.2 (1.9) | 3.0 (1.9) | 4.0 (2.8) | 3.4 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 13 | 31
  Male | 12 | 10 | 7 | 29
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Child Temperature (Degrees C)Over 6 Hours
Description: Temperature was measured hourly using a temporal thermometer to monitor the child's temperature in degrees C. Temperature of 38 degrees C or higher was considered febrile.
Time Frame: 6 hours
Population: Analysis was ITT per sample size calculation at 80% power.
Measure: Mean (Standard Deviation); unit: degrees Celcius
Arm/Group | Group A: Ibuprofen Alone | Group B: Ibuprofen and Acetaminophen | Group C: Ibuprofen Then Acetaminophen
Number analyzed (Participants) | 20 | 20 | 20
degrees Celcius | 38.5 (1.5) | 37.2 (0.6) | 36.9 (0.3)
Statistical Analysis 1: Comparison: Group A: Ibuprofen Alone vs Group B: Ibuprofen and Acetaminophen vs Group C: Ibuprofen Then Acetaminophen; Power for 80%; Test type: Non-Inferiority or Equivalence — Power for 80%; p < 0.001, Mixed Models Analysis — comparision of mean temperatures from repeated exposure. At hour 6 temperature
Statistical Analysis 2: Comparison: Group A: Ibuprofen Alone vs Group B: Ibuprofen and Acetaminophen vs Group C: Ibuprofen Then Acetaminophen; Test type: Superiority or Other; p < .0001, Chi-squared — Binary outcome <38C and >=38C

ADVERSE EVENTS:
Time Frame: 6 hours
Arm/Group | Group A: Ibuprofen Alone | Group B: Ibuprofen and Acetaminophen | Group C: Ibuprofen Then Acetaminophen
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
Relatively small sample size. Underpowered to evaluate effect oon discomfort and pain. The 6 hour observation allowed for evaluation of single cycle of drug. Did not evaluate the effect of multiple doses over a longer observation period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No